CLINICAL TRIAL: NCT06248216
Title: Implementation of an At-Home Multimodal Integrative Therapy Via Virtual Reality for Patients With Cancer-Treatment Associated Symptoms
Brief Title: Virtual Reality Therapy for Cancer-Treatment Associated Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00108489
Record Dates: First submitted 2024-01-18; First posted 2024-02-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Cancer Pain; Virtual Reality
MeSH Terms: conditions — Neoplasms; Cancer Pain

STUDY DESIGN:
Intervention Model Description: This will be a 10-week crossover design where the participants will undergo one intervention for five weeks and the other intervention for the other five weeks. Participants will be randomly assigned the order of interventions they will undergo.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study coordinator will not be blinded as they will need to administer consents and interact with participants. However, lead study investigators and outcomes assessors will be blinded to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual reality arm (Experimental): In the virtual reality intervention, participants will complete the scheduled educational module five times in the week of the intervention. This VR is assisting users in using immersive reality to reduce pain, learning cognitive and behavior self-coping skills and retraining the pain pathways. There are several sessions, which will be delivered using an all-in-one head-mounted display. Each session varies in duration approximately from 3 to 15 minutes.
  Interventions: Device: Relievrx
- Audio Mp4 arm (Placebo Comparator): In the audio intervention, participants will complete the scheduled module 5 times a week of the intervention. The content is similar to that of the VR, which will be delivered by the audio player. Each session varies in duration approximately from 3 to 15 minutes.
  Interventions: Other: Audio Mp4

INTERVENTIONS:
Device: Relievrx — The RelieVRx program is a prescription-use immersive virtual reality system intended to provide adjunctive treatment based on cognitive behavioral therapy skills and other evidence-based behavioral methods for patients (age 18 and older) with a diagnosis of chronic lower back pain (defined as moderate to severe pain lasting longer than three months). The device is intended for in-home use for the reduction of pain and pain interference associated with chronic lower back pain.
  Arms: Virtual reality arm
Other: Audio Mp4 — Audio Mp4 modules ranging from 3-15 minutes with guided meditation.
  Arms: Audio Mp4 arm

SUMMARY:
We propose an innovative approach to symptom management in cancer patients following cancer treatments, utilizing a Multimodal Integrative Therapy (MIT) delivered via Virtual Reality (VR) program, authorized by the US Food and Drug Administration for in-home use. Our primary goal is to generate pilot data on the effects of MIT-VR program on pain, fatigue, sleep, depression, and anxiety in participants suffering from chronic cancer symptoms following cancer treatments.

DETAILED DESCRIPTION:
All of the study procedures will be completed over ten weeks, during which participants will complete one in-person enrollment visit per intervention and check in-phone calls as needed during the duration of each intervention. Participants will be randomly assigned in a 1:1 fashion to one of two different interventions first: virtual reality or Mp4 audio. At home, participants will engage in their assigned intervention 5x throughout the week for five weeks using the provided device and fill out required questionnaires. Once participants complete their first intervention, they will begin the second intervention.

In the virtual reality intervention, participants will complete the scheduled educational module five times in each of the five weeks. This VR is assisting users in using immersive reality to reduce pain, learning cognitive and behavior self-coping skills and retraining the pain pathways. There are several sessions, which will be delivered using an all-in-one head-mounted display. Each session varies in duration approximately from 3 to 15 minutes. Similarly, in the audio intervention, participants will complete the scheduled module 5 times a week in each of the five weeks of the intervention. The content is similar to that of the VR, which will be delivered by the audio player. Each session varies in duration approximately from 3 to 15 minutes.

The first visit is an enrollment visit. For the enrollment visit, the participant will first complete a battery of baseline surveys. They will also receive instructions about the intervention and go through the first module of the intervention to which he or she is assigned. A member of the research team will stay with the participant while the participant completes the module to ensure the proper functioning of the device and will answer any questions that may arise. The team member will also guide the participant on how to use the device. During the five weeks of the intervention, each participant can have check-in phone calls as needed. During these check-ins, we will address any questions and issues that arise for participants to encourage compliance. Participants will return the devices after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-88
* Cancer diagnosis (histology verified)
* Had surgical intervention, completed chemotherapy or radiation for therapeutic purposes

  ->3 months since last cancer treatment, but participants currently undergoing endocrine or immunotherapy treatments are permissible
* Documented symptoms of cancer or cancer therapy including at least one of the following: pain, anxiety, sleep difficulty, fatigue, neuropathy
* English speaker (written and spoken)

Exclusion Criteria:

* Severe psychiatric condition (e.g. schizophrenia, bipolar disorders, autism) leading to hospitalization within the last 3 years
* Any personal (or family first degree) history of mania, schizophrenia, or other psychoses
* Diagnosis and treatment of chronic pain, neuropathy, fatigue, sleep or anxiety disorder prior to cancer diagnosis
* Current Hospice or palliative care only recipients
* Color-blindness
* Impaired or uncorrected hearing
* Lifetime alcohol/drug dependence or alcohol/drug abuse in past 3 months
* Conditions that would interfere with the VR mask placement (e.g. trauma, burn, infection)
* Known history of severe motion sickness
* Pregnancy or breast feeding

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
VR effect on perceived pain | Baseline to end of intervention (4 weeks)
  During daily intervention sessions (VR), participants will be required to do a pre-intervention and post-intervention survey regarding their pain (REDCAP visual analog pain survey). The post-surveys will be compared to the pre-surveys to determine VR's effect on participant pain. The surveys incorporate the Visual Analogue Scale (VAS) from 0-100, 0 being no pain experienced and 100 being the most pain experienced.
VR effect on perceived fatigue | Baseline to end of intervention (4 weeks)
  Participants will take the Patient-Reported Outcomes Measurement Information System (PROMIS) fatigue prior to intervention, and weekly throughout 4 week study period. Each follow-up survey will be compared to the baseline survey to determine VR's effect on participant fatigue. The PROMIS fatigue scale ranges from 0-50, 0 being no fatigue and 50 meaning the most fatigue.
VR effect on perceived anxiety | Baseline to end of intervention (4 weeks)
  Participants will take the PROMIS anxiety prior to intervention, and weekly throughout 4 week study period. Each follow-up survey will be compared to the baseline survey to determine VR's effect on participant anxiety. The PROMIS anxiety scale ranges from 7-35, 7 being the least anxious and 35 being the most anxious.
Audio effect on perceived pain | Baseline to end of intervention (4 weeks)
  During daily intervention sessions (audio), participants will be required to do a pre-intervention and post-intervention survey regarding their pain (REDCAP visual analog pain survey). The post-surveys will be compared to the pre-surveys to determine audio MP4's effect on participant pain. The surveys incorporate the Visual Analogue Scale (VAS) from 0-100, 0 being no pain experienced and 100 being the most pain experienced.
Audio effect on perceived fatigue | Baseline to end of intervention (4 weeks)
  Participants will take the PROMIS fatigue prior to intervention, and weekly throughout 4 week study period. Each follow-up survey will be compared to the baseline survey to determine audio MP4's effect on participant fatigue. The PROMIS fatigue scale ranges from 0-50, 0 being no fatigue and 50 meaning the most fatigue.
Audio effect on perceived anxiety | Baseline to end of intervention (4 weeks)
  Participants will take the PROMIS anxiety prior to intervention, and weekly throughout 4 week study period. Each follow-up survey will be compared to the baseline survey to determine audio MP4's effect on participant anxiety. The PROMIS anxiety scale ranges from 7-35, 7 being the least anxious and 35 being the most anxious.
Difference in effect of VR vs audio MP4 intervention on pain | Baseline to end of intervention (4 weeks)
  Scores from the daily pre and post pain surveys of each group with be compared to examine whether audio or VR had a greater impact on pain. The surveys incorporate the Visual Analogue Scale (VAS) from 0-100, 0 being no pain experienced and 100 being the most pain experienced.
Difference in effect of VR vs audio MP4 intervention on fatigue | Baseline to end of intervention (4 weeks)
  Scores from the baseline and weekly PROMIS fatigue surveys will be compared between VR and audio MP4 groups to determine if there was a differential effect on fatigue. The PROMIS fatigue scale ranges from 0-50, 0 being no fatigue and 50 meaning the most fatigue.
Difference in effect of VR vs audio MP4 intervention on anxiety | Baseline to end of intervention (4 weeks)
  Scores from the baseline and weekly PROMIS anxiety surveys will be compared between VR and audio MP4 groups to determine if there was a differential effect on anxiety. The PROMIS anxiety scale ranges from 7-35, 7 being the least anxious and 35 being the most anxious.
VR effect on perceived depression | Baseline to end of intervention (4 weeks)
  Participants will take the PROMIS depression prior to intervention, and weekly throughout 4 week study period. Each follow-up survey will be compared to the baseline survey to determine VR's effect on participant depression. The PROMIS depression scale ranges from 4-20, 4 being the least depressed and 20 being the most depressed.
Audio effect on perceived depression | Baseline to end of intervention (4 weeks)
  Participants will take the PROMIS depression prior to intervention, and weekly throughout 4 week study period. Each follow-up survey will be compared to the baseline survey to determine audio MP4's effect on participant depression. The PROMIS depression scale ranges from 4-20, 4 being the least depressed and 20 being the most depressed.
Difference in effect of VR vs audio MP4 intervention on depression | Baseline to end of intervention (4 weeks)
  Scores from the baseline and weekly PROMIS depression surveys will be compared between VR and audio MP4 groups to determine if there was a differential effect on depression. The PROMIS depression scale ranges from 4-20, 4 being the least depressed and 20 being the most depressed.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Luana Colloca, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brea-Gomez B, Torres-Sanchez I, Ortiz-Rubio A, Calvache-Mateo A, Cabrera-Martos I, Lopez-Lopez L, Valenza MC. Virtual Reality in the Treatment of Adults with Chronic Low Back Pain: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Int J Environ Res Public Health. 2021 Nov 11;18(22):11806. doi: 10.3390/ijerph182211806. PMID 34831562
- [Background] Grassini S. Virtual Reality Assisted Non-Pharmacological Treatments in Chronic Pain Management: A Systematic Review and Quantitative Meta-Analysis. Int J Environ Res Public Health. 2022 Mar 29;19(7):4071. doi: 10.3390/ijerph19074071. PMID 35409751
- [Background] Tas FQ, van Eijk CAM, Staals LM, Legerstee JS, Dierckx B. Virtual reality in pediatrics, effects on pain and anxiety: A systematic review and meta-analysis update. Paediatr Anaesth. 2022 Dec;32(12):1292-1304. doi: 10.1111/pan.14546. Epub 2022 Sep 1. PMID 35993398
- [Background] Bedford T, Adediran T, Haycock NR, Mullins CD, Medeiros M, Wright T, Curatolo M, Hamlin L, Colloca L. Patient and Provider Acceptability of a Patient Preauthorized Concealed Opioid Reduction. Pain Med. 2021 Jul 25;22(7):1651-1659. doi: 10.1093/pm/pnaa454. PMID 33674821
- [Background] Darnall BD, Krishnamurthy P, Tsuei J, Minor JD. Self-Administered Skills-Based Virtual Reality Intervention for Chronic Pain: Randomized Controlled Pilot Study. JMIR Form Res. 2020 Jul 7;4(7):e17293. doi: 10.2196/17293. PMID 32374272
- [Background] Garcia LM, Darnall BD, Krishnamurthy P, Mackey IG, Sackman J, Louis RG, Maddox T, Birckhead BJ. Self-Administered Behavioral Skills-Based At-Home Virtual Reality Therapy for Chronic Low Back Pain: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jan 19;10(1):e25291. doi: 10.2196/25291. PMID 33464215
- [Background] Garcia LM, Birckhead BJ, Krishnamurthy P, Sackman J, Mackey IG, Louis RG, Salmasi V, Maddox T, Darnall BD. An 8-Week Self-Administered At-Home Behavioral Skills-Based Virtual Reality Program for Chronic Low Back Pain: Double-Blind, Randomized, Placebo-Controlled Trial Conducted During COVID-19. J Med Internet Res. 2021 Feb 22;23(2):e26292. doi: 10.2196/26292. PMID 33484240
- [Background] Garcia LM, Birckhead BJ, Krishnamurthy P, Mackey I, Sackman J, Salmasi V, Louis R, Maddox T, Darnall BD. Three-Month Follow-Up Results of a Double-Blind, Randomized Placebo-Controlled Trial of 8-Week Self-Administered At-Home Behavioral Skills-Based Virtual Reality (VR) for Chronic Low Back Pain. J Pain. 2022 May;23(5):822-840. doi: 10.1016/j.jpain.2021.12.002. Epub 2021 Dec 11. PMID 34902548
- [Background] Garcia L, Birckhead B, Krishnamurthy P, Mackey I, Sackman J, Salmasi V, Louis R, Castro C, Maddox R, Maddox T, Darnall BD. Durability of the Treatment Effects of an 8-Week Self-administered Home-Based Virtual Reality Program for Chronic Low Back Pain: 6-Month Follow-up Study of a Randomized Clinical Trial. J Med Internet Res. 2022 May 25;24(5):e37480. doi: 10.2196/37480. PMID 35612905
- [Background] Maddox T, Sparks C, Oldstone L, Maddox R, Ffrench K, Garcia H, Krishnamurthy P, Okhotin D, Garcia LM, Birckhead BJ, Sackman J, Mackey I, Louis R, Salmasi V, Oyao A, Darnall BD. Durable chronic low back pain reductions up to 24 months after treatment for an accessible, 8-week, in-home behavioral skills-based virtual reality program: a randomized controlled trial. Pain Med. 2023 Oct 3;24(10):1200-1203. doi: 10.1093/pm/pnad070. No abstract available. PMID 37220894
- [Background] Kelleher SA, Fisher HM, Winger JG, Miller SN, Amaden GH, Somers TJ, Colloca L, Uronis HE, Keefe FJ. Virtual reality for improving pain and pain-related symptoms in patients with advanced stage colorectal cancer: A pilot trial to test feasibility and acceptability. Palliat Support Care. 2022 Aug;20(4):471-481. doi: 10.1017/S1478951521002017. PMID 35078545
- [Result] Zeng Y, Zhang JE, Cheng ASK, Cheng H, Wefel JS. Meta-Analysis of the Efficacy of Virtual Reality-Based Interventions in Cancer-Related Symptom Management. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419871108. doi: 10.1177/1534735419871108. PMID 31441352